CLINICAL TRIAL: NCT00977977
Title: Rituximab Plus Cyclosporine in Idiopathic Membranous Nephropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090223; 09-DK-0223
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-08-04

CONDITIONS: Nephrotic Syndrome; Proteinuria; Autoimmune Disease; Glomerular Disease; Membranous Glomerulonephritis
Keywords: Kidney Disease; Nephrotic Syndrome; Autoimmune Diseases; Clinical Trial; Proteinuria
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria; Autoimmune Diseases; Glomerulonephritis, Membranous; Kidney Diseases | interventions — Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of Rituximab plus cyclosporine (Experimental): 2 infusions (each 1000 mg) separated by 2 weeks; repeated after 6 months. Daily therapy for 6 months (3-5 mg/kg), then tapered and discontinued.
  Interventions: Drug: Rituximab Infusion; Drug: Oral Cyclosporine

INTERVENTIONS:
Drug: Rituximab Infusion — Drug Rituximab Infusion 2 infusions (each 1000 mg) separated by 2 weeks; repeated after 6 months
Drug: Oral Cyclosporine — Daily therapy for 6 months (3-5 mg/kg), then tapered and discontinued

SUMMARY:
Background:

* Membranous nephropathy is associated with damage to the walls of the glomeruli, the small blood vessels in the kidneys that filter waste products from the blood. This damage causes leakage of blood proteins into the urine and is associated with low blood protein levels, high blood cholesterol values, and swelling of the legs. These problems can decrease or go away without treatment in about 25 percent of patients, but if they persist, some patients may experience impaired (or loss of) kidney function, blood vessel and heart disease, and a risk of forming blood clots in veins.
* Kidney biopsies that show that antibodies have been deposited along the glomeruli suggest that specialized cells of the immune system, called B and T cells, are causing damage to the kidneys through their increased activity. To suppress the action of B and T cells and to decrease the harmful deposits in the kidneys, drug treatments are required.
* Patients with membranous nephropathy are often treated with immunosuppressive drugs such as cyclosporine or cytoxan plus steroids that attempt to reduce or suppress the activity of the immune system, decrease antibody production, and reduce antibody deposits in the kidney. However, not everyone responds to these medications and the kidney disease can return in some patients when the drugs are stopped. Also, there are side effects associated with long term usage of these medications. Rituximab, a different immunosuppressant, has also been used for this purpose. Although cyclosporine and Rituximab have been used separately, they have not been tried in combination as a possible treatment for membranous nephropathy.

Objectives:

- To determine the safety and effectiveness of combining rituximab and cyclosporine to treat membranous nephropathy.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with membranous nephropathy based on a kidney biopsy done within the preceding 24 months, and who have had excess levels of protein in the urine for at least 6 months based on urine and blood tests.

Design:

* Potential participants will be screened with an initial clinic evaluation and full medical history.
* Before the treatment, there will be a run-in period that will last up to 2 months. During this time, participants will be placed on a blood pressure lowering medication and will not take any other immunosuppressant medications.
* Participants will visit the NIH clinical center for a baseline evaluation, four intravenous infusions of rituximab, and also at 1- to 6-month intervals throughout the study.
* Active treatment period will involve a 6-month course of cyclosporine and a total of four doses of rituximab. Participants will take cyclosporine tablets twice daily, and have two infusions of rituximab given 2 weeks apart, After 6 months, the cyclosporine dose will slowly be decreased over several weeks and then completely discontinued. Participants will then receive another course (two doses 2 weeks apart) of rituximab, depending on results of blood work.
* Participants will have frequent blood and urine tests performed to monitor the results of treatment and reduce the chance of side effects.

DETAILED DESCRIPTION:
Study Description:

Subjects with idiopathic membranous nephropathy will be treated with a combination of rituximab and cyclosporine. The study hypothesis of combining Rituximab and cyclosporine provides more effective immunosuppression than either agent alone by targeting both arms of the immune system which are believed to be involved in the pathogenesis of MN. The combination of Rituximab and cyclosporine may achieve greater reductions in proteinuria, increase the number of remissions (especially complete) of the nephrotic syndrome, decrease the number of relapses and perhaps reset the immune system, thereby obviating the need for long term immunosuppression. The prolonged effects of Rituximab on the immune system may allow for withdrawal of cyclosporine. Although each of these medications has been used separately in membranous nephropathy, the potential benefits and risks of this combination have not yet been formally explored.

Objectives:

Primary objective:

To determine the safety and effectiveness of combining rituximab and cyclosporine to treat membranous nephropathy by evaluating the acceptable safety profile and efficacy to reduce proteinuria.

Secondary objective:

To evaluate the efficacy to maintain durable remission.

Endpoints:

Primary endpoint:

Incidence of adverse events (AEs) will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE).

Number of subjects who achieve complete remission (CR), partial remission (PR) at 6, 12, and 18 months.

Secondary endpoint:

1. Time to remission
2. Time to relapse (in those who achieved a remission)
3. Change in proteinuria from baseline to 12 months

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, >= 18 years of age
3. Nephrotic range proteinuria that persists for at least 6 months post diagnosis of membranous nephropathy greater than 3.5 grams /24 hours (based on 24-hour urine collection).

   a. If the subject s renal function rapidly declines in less than 6 months could proceed with immunosuppression therapy sooner such as complications of the nephrotic syndrome that are not controlled with supportive therapy or evidence of decline in glomerular filtration rate or proteinuria >8 grams/day. Subjects with declining renal function and/or high-grade proteinuria due to MN are considered "high risk" subjects and have a higher probability of progression to end stage kidney disease.
4. Nephrotic range proteinuria (>3.5 g/24 hours) that persists despite angiotensin antagonist therapy (ACE inhibitor or ARB) for at least 2 months unless intolerant.

   a. The rationale is that blockade of the renin angiotensin system (RAAS) is widely considered to be part of the standard of care treatment for subjects with the nephrotic syndrome. Nephrotic range proteinuria will be defined as an estimated average proteinuria >3.5 g/24 hours in adults based on at least two 24-hour urine protein excretions obtained prior to initiating therapy. Incomplete urine

   collections (based on inadequate creatinine excretion) will be excluded.
5. Renal biopsy within the past 24 months must reveal typical changes of membranous nephropathy by light and electron microscopy or a positive anti-PLA2R antibody test in the serum. There has been a change in the management strategies for MN such that a renal biopsy is not absolutely required for diagnosis if patient has positive circulating anti-PLA2R antibody.

   a. Based on published KDIGO 2021 Clinical Practice Guidelines 3.1.1 patients with MN who are positive for anti-PLA2R do not require renal biopsy as long as renal function is normal (eGFR >60) and has not had immunosuppression as it has been demonstrated that results of the biopsy have not altered clinical approach and management. If not PLA2R positive, renal biopsy within 24 months is still required.
6. Blood pressure <=140/90 on >75% of measurement while on anti-hypertensive treatment for at least 1-2 months.
7. There is no evidence to suggest secondary forms of membranous nephropathy.
8. Ability to take oral medication and be willing to adhere to the cyclosporine regimen
9. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for 12 months after the last Rituximab infusion.
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
11. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Estimated GFR<40 ml/min/1.73 m^2 from the preceding 2 months prior to enrollment while on ACEI/ARB therapy.
2. Immunosuppressive medications or experimental medications of any type during the three-month period prior to initiating Rituximab and cyclosporine.
3. Prior exposure to cyclosporine or tacrolimus for more than 6 months and/or evidence of intolerance or toxicity associated with cyclosporine treatment of any duration including irreversible azotemia, liver dysfunction or hypertension
4. Rituximab use within the previous 12 months.
5. Clinically significant medical conditions (i.e., severe heart failure NYHA class IV, uncontrolled coronary artery disease/unstable angina), which in the opinion of the investigator, could increase the subject s risk of participating in the study or could confound the interpretation of the results of the study.
6. Positive HIV serology
7. Positive HCV serology
8. Active acute or chronic infection requiring antimicrobial therapy or serious viral infection cytomegalovirus, herpes simplex, varicella zoster virus (chicken pox or shingles), Parvovirus B19 (can be based on previous medical records within the past 24-months)
9. Live viral vaccines within one month prior to Rituximab.
10. Pregnancy or lactation
11. Cancer diagnosis or cancer recurrence within the preceding 5 years, excluding basal cell carcinoma of the skin. The rationale is that immunosuppression may accelerate cancer progression.
12. Clinical evidence of cirrhosis or chronic active liver disease sufficiently severe to impair cyclosporine metabolism; this would include a prolonged prothrombin time.
13. Cytopenia (neutrophils <1500/mm^3 and/or thrombocytopenia <75,000) and/or CD4 T cell count <200/mm^3). The rationale is that Rituximab therapy may be followed by cytopenia with the granulocyte lineage being at greatest risk. Patients with low CD4 T cell counts are prone to infection which can be exacerbated by Rituximab.
14. Diabetes mellitus. The rationale is that diabetes may lead to worsening of proteinuria that would not respond to immunosuppression and would confound the results.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 24 months
  Safety 24 months We will assess using the National Cancer Institute common Terminology Criteria for Adverse Events (CTCAE)
Percentage of complete and partial remissions (CR and PR) | 6 months
  Proteinuria; complete remission (CR) defined as less than 300 mg/24 proteinuria and partial remission (PR) <3.5 grams/day and >=50%reduction of proteinuria
Percentage of complete and partial remissions (CR and PR) | 24 months
  Proteinuria; complete remission (CR) defined as less than 300 mg/24 proteinuria and partial remission (PR) <3.5 grams/day and >=50%reduction of proteinuria
Percentage of complete and partial remissions (CR and PR) | 18 months
  Proteinuria; complete remission (CR) defined as less than 300 mg/24 proteinuria and partial remission (PR) <3.5 grams/day and >=50%reduction of proteinuria
Percentage of complete and partial remissions (CR and PR) | 12 months
  Proteinuria; complete remission (CR) defined as less than 300 mg/24 proteinuria and partial remission (PR) <3.5 grams/day and >=50%reduction of proteinuria

SECONDARY OUTCOMES:
Time to remission Baseline to 24 months | Baseline to 24 months
Time to relapse (in those who achieved a remission) | Baseline to 24 months
Change in proteinuria from baseline to 12 months | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Meryl A Waldman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - National Naval Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glassock RJ. Diagnosis and natural course of membranous nephropathy. Semin Nephrol. 2003 Jul;23(4):324-32. doi: 10.1016/s0270-9295(03)00049-4. PMID 12923720
- [Background] Cattran D. Management of membranous nephropathy: when and what for treatment. J Am Soc Nephrol. 2005 May;16(5):1188-94. doi: 10.1681/ASN.2005010028. Epub 2005 Mar 30. No abstract available. PMID 15800117
- [Background] Kerjaschki D, Neale TJ. Molecular mechanisms of glomerular injury in rat experimental membranous nephropathy (Heymann nephritis). J Am Soc Nephrol. 1996 Dec;7(12):2518-26. doi: 10.1681/ASN.V7122518. PMID 8989729
- [Derived] Burbelo PD, Olson SW, Keller JM, Joshi M, Schwartz DM, Chuang YJ, Lambeau G, Beck LH Jr, Waldman M. Prediagnostic Appearance of Thrombospondin Type-1 Domain 7A Autoantibodies in Membranous Nephropathy. Kidney360. 2023 Feb 1;4(2):217-225. doi: 10.34067/KID.0005112022. Epub 2022 Nov 29. PMID 36821613
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-DK-0223.html